CLINICAL TRIAL: NCT05736029
Title: PROPHETIC Extended - Predicting Responsiveness in Oncology Patients Based on Host Response Evaluation During Anti Cancer Treatments, Extended Study.
Brief Title: Predicting Responsiveness in Oncology Patients Based on Host Response Evaluation During Anti Cancer Treatments, Using Multiomics
Acronym: PROPHETIC
Status: Recruiting | Type: Observational
Sponsor: OncoHost Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OH-HRPP-002
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Non Small Cell Lung Cancer; Healthy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. plasma samples
  2. PBMCs
  3. Stool samples
  4. Tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-operable NSCLC patients receiving ICI therapy: Patients with non-operable stage IIIB-IV NSCLC treated with immune check inhibitor anti cancer treatment as a standard of care
  Interventions: Other: blood, stool and tissue samples collection
- Operable NSCLC Patients Receiving ICI as Neoadjuvant or Adjuvant Therapy: Patients with operable stage II-IIIA NSCLC, treated with immune check inhibitor in the neoadjuvant or adjuvant setting
  Interventions: Other: blood, stool and tissue samples collection
- Healthy volunteers: Sex and aged matched non-diseased volunteers
  Interventions: Other: blood, stool and tissue samples collection

INTERVENTIONS:
Other: blood, stool and tissue samples collection — blood, stool and tissue samples collection before and during the treatment, as applicable

SUMMARY:
The goal of this exploratory study is understand the mechanisms of response to immunotherapy in Non-Small Cell Lung Cancer patients.

The investigators are going to search for correlation between specific biological features and response to immunotherapy, and to use those associations for developing an algorithm enabling to identify patients that could benefit from the immune check inhibitor based anti cancer treatment.

Patients will provide biological samples before and during their treatment, and clinical data will be collected.

DETAILED DESCRIPTION:
The goal of the study is to develop an algorithm that associates between biomarkers detected in biospecimen of NSCLC patients, and their:

* Response to treatment
* Clinical benefit parameters such as PFS and OS.
* Adverse events to immune check inhibitor therapy
* Biological mechanisms involved in response or resistance to immune check inhibitor therapy.

Patients will provide plasma, PBMCs, stool and tissue samples (where applicable) before and during treatment.

Clinical data, including disease history, given treatment, response evaluation and adverse events to the treatment will be recorded.

Samples will be analysed as follows -

* Proteomic features (Plasma proteomics)
* Epigenetic patterns (cell free DNA)
* ctDNA mutation analysis
* PBMC subpopulations
* Microbiome profiling (Stool)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures.
* Male or female aged at least 18 years.
* ECOG PS - 0/1-2.

Exclusion Criteria:

* Any concurrent and/or other active malignancy that has required systemic treatment within 2 years of first dose of treatment.
* Generalized impairment or mental incompetence that would render the patient unable to understand his/her participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population comprises 3 sub-populations:
  Cohort 1 - Non-operable NSCLC (Stages IIIB to IV), receiving immune-check inhibitor (ICI) therapy [any combination of ICI / ICI ±Chemotherapy, and any line of treatment].
  Cohort 2 - Operable NSCLC (Stages II-IIIA), receiving ICI in the neoadjuvant or adjuvant setting.
  Cohort 3 - Sex and aged matched non-diseased volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response (OR) | month 3
  OR as defined by RECIST 1.1 or any other validated clinical scale for response
Overall response (OR) | month 6
  OR as defined by RECIST 1.1 or any other validated clinical scale for response
Overall response (OR) | month 9
  OR as defined by RECIST 1.1 or any other validated clinical scale for response
Overall response (OR) | month 12
  OR as defined by RECIST 1.1 or any other validated clinical scale for response
Overall response (OR) | month 15
  OR as defined by RECIST 1.1 or any other validated clinical scale for response
Overall response (OR) | month 18
  OR as defined by RECIST 1.1 or any other validated clinical scale for response
Overall response (OR) | month 21
  OR as defined by RECIST 1.1 or any other validated clinical scale for response
Overall response (OR) | month 24
  OR as defined by RECIST 1.1 or any other validated clinical scale for response
Plasma proteomic profile | Baseline, pre treatment
  Plasma proteins measurments
Plasma proteomic profile | 2(+/-1) weeks from first treatment
  Plasma proteins measurments
Plasma proteomic profile | 3 months
  Plasma proteins measurments
Plasma proteomic profile | 6 months
  Plasma proteins measurments
Plasma proteomic profile | 9 months
  Plasma proteins measurments
Plasma proteomic profile | 12 months
  Plasma proteins measurments
Plasma proteomic profile | 15 months
  Plasma proteins measurments
Plasma proteomic profile | 18 months
  Plasma proteins measurments
Plasma proteomic profile | 21 months
  Plasma proteins measurments
Plasma proteomic profile | 24 months
  Plasma proteins measurments
Epigenetic patterns | Baseline, pre treatment
  Characterization of Cell free DNA
Epigenetic patterns | 2(+/-1) weeks from first treatment
  Characterization of Cell free DNA
Epigenetic patterns | 12 months
  Characterization of Cell free DNA
Epigenetic patterns | 24 months
  Characterization of Cell free DNA
ctDNA mutation analysis | immediately after surgery
  ctDNA mutation analysis
Microbiome profiling | Baseline, pre treatment
  PBMC subpopulations exploration
Microbiome profiling | 2(+/-1) weeks from first treatment
  PBMC subpopulations exploration
Microbiome profiling | 12 months
  PBMC subpopulations exploration
Microbiome profiling | 24 months
  PBMC subpopulations exploration

OTHER OUTCOMES:
Progression Free Survival (PFS) | From date of enrollment until the date of first documented progression, assessed up to 100 months
  Documentation of Progression Free Survival (PFS) duration
Overall Survival (OS) | From date of enrollment until the date of death from any cause, assessed up to 100 month
  Documentaion of Overall Survival (OS) duration
Adverse Events (AE) | 3 months
  AE, as reported by the patients
Adverse Events (AE) | 6 months
  AE, as reported by the patients
Adverse Events (AE) | 9 months
  AE, as reported by the patients
Adverse Events (AE) | 12 months
  AE, as reported by the patients
Adverse Events (AE) | 15 monthst
  AE, as reported by the patients
Adverse Events (AE) | 18 months
  AE, as reported by the patients
Adverse Events (AE) | 21 months
  AE, as reported by the patients
Adverse Events (AE) | 24 months
  AE, as reported by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Ronan J Kelly, MD MBA, Principal Investigator — Chief of Oncology Baylor Scott & White Health System
Locations (1):
- Baylor Scott and White Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No